CLINICAL TRIAL: NCT02685696
Title: To Investigate the Incidence of Surgical Site Infection in Low Risk Women Having a First Time Planned Caesarean Section Using the Alexis O Retractor and the Traditional Metal Retractor
Brief Title: Surgical Site Infection in Caesarean Section Using Alexis O Compared to Metal Retractors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Larry Hinkson, Consultant in Obstetrics, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AlexisO1
Record Dates: First submitted 2016-02-08; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alexis O Retractor (Experimental): Group 1 received the Alexis-O-Retractor at thet time of first Caesarean Section
  Interventions: Device: Alexis O Retractor
- Metal Retractor (Active Comparator): Group 2 received the traditional self retaining metal Retractor at thet time of first Caesarean Section
  Interventions: Device: Metal Retractor

INTERVENTIONS:
Device: Alexis O Retractor — A newly developed abdominal wall retractor for Caesarean Section is the Alexis O Ring which is formed of 2 rings and a interconnecting plastic polyurethane sheath where the flexible inner ring is placed into the abdomen and where the rigid outer ring is rolled to create tension on the plastic sheath providing 360° abdominal wound retraction with simultaneously a tamponade effect whilst covering the abdominal wound during the Caesarean Section and delivery of the baby.
  Arms: Alexis O Retractor
Device: Metal Retractor — The traditional self-retaining metal Collins Caesarean Wound Retractor.
  Other Names: Collins
  Arms: Metal Retractor

SUMMARY:
Objective:

To investigate if the use of the newly designed Alexis O Retractor leads to improved intra-operative and post-operative surgical outcomes in the setting of planned elective Caesarean Sections.

Study Design:

This ethically approved study is designed as a prospective, randomized controlled trial in planned, first time Caesarean Sections with 200 patients randomized to either the Alexis-O Retractor group or the conventional group. Patients with wound healing problems, connective tissue disorders, insulin dependent diabetes, bleeding disorders, previous major abdominal surgery and chorioamnionitis are excluded. Outcomes include surgical site infection, intraoperative parameters such as tissue damage, postoperative analgesia requirements and patient satisfaction scores.

DETAILED DESCRIPTION:
Main Hypothesis:

Does the use of the newly designed Alexis O Retractor lead to improved Surgical Site Infection rates intra-operative and post-operative surgical outcomes in the setting of planned elective first time Caesarean Sections in patients compared to the traditional self-retaining metal retractor?

Secondary Hypotheses:

Does the Alexis O Retractor lead to improved intra-operative and post-operative surgical outcomes in the setting of planned elective Caesarean Sections?

Study Design:

The Study is designed as a prospective, randomized controlled trial with 100 patients randomized to the Alexis O Retractor group and 100 patients to the conventional group.

All patients will be recruited following a thorough discussion about the purpose and methodology of the study and full documented consent will be obtained prior to randomization.

Patients with wound healing problems, connective tissue disorders, diabetes, bleeding disorders, previous abdominal surgery apart from laparoscopy and chorioamnionitis will be excluded.

All surgical operators are thoroughly trained in the use and application of the Alexis O Retractor prior to the start of the study and supported by regular teaching demonstrations. The Obstetric Theatre Team is informed and trained in use and application of the Alexis O Retractor within the Study Design.

Ethical Approval:

Ethical Approval has already been obtained from the Ethics committee at the Charité University Hospital Committee and in keeping with ethical standards.

Statistics:

* Data analysis and statistical comparisons will be performed by the appropriate robust statistical methodology.
* Comparisons to be investigated
* Subjective Assessment of the Ease of Application of Retractor Instrument
* Incision to Delivery Time
* Incision to Skin Suture Time
* Subjective Assessment of Visualized Operative Field
* Subjective Assessment of Freedom of Surgical Movement
* Interference from Descending Bowel or Adnexal Tissue
* Bowel and Bladder Trauma
* Need for Bowel Packing
* Need for Paracolic Cleaning of Blood and Amniotic Fluid
* Need for Uterus Exteriorization Intraoperatively
* Fascial Trauma
* Muscle Trauma
* Muscle Suturing
* Coagulation of the Subcutaneous Tissue
* Subcutaneous Tissue Thickness
* Skin Lacerations
* Trauma to the Baby
* Estimated Blood Loss
* Ease of Retractor Removal
* Analgesia Requirements Post Operative
* Wound Healing Problems on Discharge and at 6 Weeks (Telephone Interview)
* Wound Infections (As defined by Centers for Disease Control)
* Time to Hospital Discharge
* 6-Week Scar Pain Scores (Telephone Interview)
* Patient Satisfaction with Wound Healing (Telephone Interview)

ELIGIBILITY:
Inclusion Criteria:

* Women
* Elective Caesarean Section
* First Caesarean Section

Exclusion Criteria

* Diabetes
* Chronic auto immune diseases
* Lupus
* Immune deficiency diseases
* HIV
* known bleeding disorders
* full anti-coagulation therapy
* wound healing problems
* previous Caesarean Section
* major abdominal surgery
* laparotomy
* active phase of labor
* suspected chorioamnionitis
* confirmed chorioamnionitis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection in low risk women having a first time planned Caesarean Section using the Alexis O Retractor compared to the traditional Metal Retractor. | 6-8 Weeks after Surgery

SECONDARY OUTCOMES:
Application Satisfaction Scale Scores | Immediate Postoperative
Removal Satisfaction Scale Scores | On the day of Surgery (Day 0)
Post Operative Pain Scale Scores at Discharge | On the day of discharge (3-5 days)
Post Operative Pain at 6 Weeks | 6 weeks post operative
Patients with Wound Dehisence at Discharge | On the day of discharge (3-5 days)
Patients with either open wounds, infected wounds, bleeding wounds or painful wound at 6 Weeks | 6 weeks post operative
Blood Loss Volume | On the day of Surgery (Day 0)
Visual Field Satisfaction Scores | On the day of Surgery (Day 0)
Freedom of Movement Satisfaction Scores | On the day of Surgery (Day 0)
No. Patients with Prolapsing Bowel in the operative field at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients needing repositioning of prolapsing bowel at the time of Caesarean | On the day of Surgery (Day 0)
No. of Patients with bowel injury sustained at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients sustaining bladder injury at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients where bowel packing with abdominal swabs was performed at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients where suction of Blood and Liquor from the parabolic gutters was necessary at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients where the Uterus was exteriorized at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients with Rectus Sheath Fascial Tears at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients with Rectus Muscle Tearing at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients where Rectus Muscle Suturing was performed at the time of Caesarean | On the day of Surgery (Day 0)
No. of Patients where Subcutaneous Electro-Coagulation was performed at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients with lacerations to the skin wound edges at the time of Caesarean Section | On the day of Surgery (Day 0)
No. of Patients where the Baby was cut at the time of Caesarean Section | On the day of Surgery (Day 0)
Wound Healing Satisfaction at 6 Weeks | 6 weeks post operative.
Time to Discharge | 3-5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hinkson, MBBS,MRCOG, Principal Investigator — Charité University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klingel ML, Patel SV. A meta-analysis of the effect of inspired oxygen concentration on the incidence of surgical site infection following cesarean section. Int J Obstet Anesth. 2013 Apr;22(2):104-12. doi: 10.1016/j.ijoa.2013.01.001. Epub 2013 Mar 13. PMID 23490472
- [Background] Horiuchi T, Tanishima H, Tamagawa K, Sakaguchi S, Shono Y, Tsubakihara H, Tabuse K, Kinoshita Y. A wound protector shields incision sites from bacterial invasion. Surg Infect (Larchmt). 2010 Dec;11(6):501-3. doi: 10.1089/sur.2009.072. Epub 2010 Sep 17. PMID 20849290